CLINICAL TRIAL: NCT06467916
Title: The Development of PATH, a Program to Support NICU Parent Mental Health Through the Transition From Hospital to Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Oregon Health and Science University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-1191; K08MH127519 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Perinatal Mental Health
Keywords: neonatal intensive care unit; perinatal mental health; perinatal depression; perinatal anxiety; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): anticipatory guidance, brief behavioral intervention, or referral to community mental health provider
  Interventions: Behavioral: Behavioral Treatment
- Control (No Intervention): usual care

INTERVENTIONS:
Behavioral: Behavioral Treatment — anticipatory guidance, brief behavioral intervention, or referral to community mental health provider
  Arms: Intervention

SUMMARY:
The objective of this study is to develop and pilot test a telehealth-based mental health screening and engagement program that supports parents as their infants transition home from the NICU. The program will use a stepped-care approach to screen parents for depression, anxiety, and PTSD; provide a brief behavioral intervention to those who screen as having at least a low risk of these conditions; and provide a warm hand-off to community mental health services for those at medium to high risk.

ELIGIBILITY:
Inclusion Criteria:

* NICU parents: Participants will be parents of currently hospitalized preterm infants from either the OHSU NICU or the UCH NICU. We will include parents of live preterm infants who have been admitted in the NICU for at least 2 weeks. Parents must speak English or Spanish. Parents can be of any age.
* NICU stakeholders: Participants will be stakeholders from either the OHSU NICU or the UCH NICU. Stakeholders will be social workers, mental health providers responsible for providing more intensive mental health support for NICU parents, nurses, neonatologists, and hospital administrators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mental health self-efficacy scale | ~2 weeks prior to discharge; 2 weeks post-discharge; 6 weeks post-discharge
  Mental health self-efficacy

SECONDARY OUTCOMES:
City Mental Illness Stigma Scale | ~2 weeks prior to discharge; 2 weeks post-discharge; 6 weeks post-discharge
  Mental illness stigma
Parenting Sense of Self Confidence Scale | ~2 weeks prior to discharge; 2 weeks post-discharge; 6 weeks post-discharge
  Parenting self-efficacy

OTHER OUTCOMES:
Edinburgh Postnatal Depression Scale (EDPS) | ~2 weeks prior to discharge; 2 weeks post-discharge; 6 weeks post-discharge
  Perinatal depression
GAD-7 | ~2 weeks prior to discharge; 2 weeks post-discharge; 6 weeks post-discharge
  Anxiety
Post-Traumatic Stress Disorder Questionnaire (PPQ) | ~2 weeks prior to discharge; 2 weeks post-discharge; 6 weeks post-discharge
  PTSD

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Project data and materials will be administered in accordance with both participating institutional and NIH policies, including the NICH Data Sharing Policy and Implementation Guidance of March 5, 2003. Depending on such policies, materials may be transferred to others under the terms of material transfer agreement. Data, including survey instruments and datasets, will be available approximately one year after study completion. Researchers can contact the research staff to request access to datasets and support for their use. Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices. The final locked dataset will be stripped of all participant identifiers. This dataset will be available to the nonprofit community for noncommercial uses provided that a data-sharing agreement is reached and that the original creators of the dataset are able to collaborate in all secondary data analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All shareable, de-identified scientific data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 3 years after the funding period.
Access Criteria: Scientific data will be findable for the research community through PubMed Central. For all publications, a digital object identifier (DOI) will be created. The data DOI will be referenced in the publication to allow the scientific community easy access to the data used in the publication.